CLINICAL TRIAL: NCT07380035
Title: Voluntariness of Same-Day Consent for Participation in Low-Risk Clinical Anesthesia Research Trials: A Prospective, Randomized Trial
Brief Title: Coercion in Same-Day Research Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Women's College Hospital (Other); Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Connor Brenna, Resident Physician, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2023-0007-E; 46twc (Other: Open Science Framework)
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Consent of Patients; Coercion to Participate in Research
Keywords: Coercion; Voluntariness; Research consent; Clinical trials; Perioperative research

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance Consent (Sham Comparator): Patients in this group were presented with the opportunity for trial participation in advance of surgery, during preoperative assessment approximately one week prior in the Pre-Anesthesia Clinic. Recruitment took place via telephone during this pre-operative assessment, and followed all standard procedures for trial recruitment at Women's College Hospital.
  Interventions: Other: Invitation to Consent to Trial Participation
- Day of Surgery Consent (Experimental): Patients in this group were presented with the opportunity for trial participation on the day of surgery, immediately before proceeding to their operation at Women's College Hospital. Recruitment took place in person at the bedside, and otherwise followed all standard procedures for trial recruitment at Women's College Hospital.
  Interventions: Other: Invitation to Consent to Trial Participation

INTERVENTIONS:
Other: Invitation to Consent to Trial Participation — In this trial, the intervention being studied was the timing of an invitation to participate in a fabricated low-risk clinical anesthesia research trial. Patients were recruited into this fictitious trial either several days in advance of surgery, or on the day of surgery, and post-operative evaluations aimed to measure whether these groups experienced different degrees of coercion or voluntariness in their decisions to participate.

SUMMARY:
As a result of their unique practice patterns, many specialist physicians typically only meet patients on the date of an intervention such as surgery. However, some of the world's most prestigious academic centers do not allow research participants to be recruited on the same day as surgery. This is because of concerns, shared by researchers and research ethics boards, that patients may be too anxious or rushed to provide informed, voluntary consent immediately before an operation. This is not supported by evidence, and leads to potential inequities by restricting patients' opportunities to contribute to and benefit from research. The investigators undertook a randomized controlled trial incorporating deception to study the voluntariness of research consent provided by patients invited to enroll in a fabricated anesthesia research study at Women's College Hospital in Toronto, Ontario, Canada. Patients undergoing day surgery were randomized to receive research recruitment opportunities either days before surgery in the pre-operative assessment clinic, or on the surgical date. Post-operatively, patient's perceptions of undue influence or coercion in the consent process were examined with questionnaires and compared between these groups. This trial will help to design future perioperative studies, and will answer the important question of whether truly voluntary and informed same-day consent can be provided for participation in perioperative research.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo ambulatory anterior cruciate ligament repair under general anesthesia with an adductor canal nerve block at Women's Colege Hospital
* Age ≥18

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Average score on combined modified coercion scales | Measured on postoperative day one.
  Minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion.
Average Score on modified Iowa Coercion Questionnaire | Measured on postoperative day one.
  Minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion.
Average Score on Modified Coercion Assessment Scale | Measured on postoperative day one.
  Minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion.

SECONDARY OUTCOMES:
Rate of enrollment into the fictitious trial | Measured when patients were approached with an invitation to participate in the trial. For patients in the Advance Consent Group this was, on average, preoperative day seven. For patients in the Day of Surgery Group this was postoperative day zero.
Responses to individual items on the combined modified coercion scales | Measured on postoperative day one.
  Each item has a minimum score of 1 and maximum score of 4, with higher scores corresponding to a greater degree of coercion.

OTHER OUTCOMES:
Association between participant sex and average score on combined modified coercion scales | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant sex (categorical variable self-reported on the postoperative questionnaire) and average score on the combined modified coercion scales (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant sex and average score on the modified Iowa Coercion Questionnaire | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant sex (categorical variable self-reported on the postoperative questionnaire) and average score on the modified Iowa Coercion Questionnaire (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant sex and average score on the modified Coercion Assessment Scale | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant sex (categorical variable self-reported on the postoperative questionnaire) and average score on the modified Coercion Assessment Scale (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant age and average score on combined modified coercion scales | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant age (continuous variable self-reported on the postoperative questionnaire) and average score on the combined modified coercion scales (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant age and average score on the modified Iowa Coercion Questionnaire | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant age (continuous variable self-reported on the postoperative questionnaire) and average score on the modified Iowa Coercion Questionnaire (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant age and average score on the modified Coercion Assessment Scale | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant age (continuous variable self-reported on the postoperative questionnaire) and average score on the modified Coercion Assessment Scale (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant education and average score on combined modified coercion scales | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant total years of education (continuous variable self-reported on the postoperative questionnaire) and average score on the combined modified coercion scales (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant education and average score on the modified Iowa Coercion Questionnaire | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant total years of education (continuous variable self-reported on the postoperative questionnaire) and average score on the modified Iowa Coercion Questionnaire (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant education and average score on the modified Coercion Assessment Scale | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant total years of education (continuous variable self-reported on the postoperative questionnaire) and average score on the modified Coercion Assessment Scale (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant country of upbringing and average score on combined modified coercion scales | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant country of upbringing (categorical variable self-reported on the postoperative questionnaire) and average score on the combined modified coercion scales (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant country of upbringing and average score on the modified Iowa Coercion Questionnaire | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant country of upbringing (categorical variable self-reported on the postoperative questionnaire) and average score on the modified Iowa Coercion Questionnaire (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant country of upbringing and average score on the modified Coercion Assessment Scale | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant country of upbringing (categorical variable self-reported on the postoperative questionnaire) and average score on the modified Coercion Assessment Scale (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant minority status and average score on combined modified coercion scales | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant minority status (categorical variable self-reported on the postoperative questionnaire) and average score on the combined modified coercion scales (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant minority status and average score on the modified Iowa Coercion Questionnaire | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant minority status (categorical variable self-reported on the postoperative questionnaire) and average score on the modified Iowa Coercion Questionnaire (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).
Association between participant minority status and average score on the modified Coercion Assessment Scale | Measured on postoperative day one.
  This secondary analysis uses linear regression to test for statistical dependence between participant minority status (categorical variable self-reported on the postoperative questionnaire) and average score on the modified Coercion Assessment Scale (minimum average score of 1 and maximum average score of 4, with higher scores corresponding to a greater degree of coercion).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, aggregate trial data supporting the findings of this study will be made available upon reasonable request to the corresponding author after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Brenna CTA, Walton N, Cohn M, Siddiqui U, Huszti E, Brull R. Coerced consent in clinical research: study protocol for a randomized controlled trial. Trials. 2024 Jul 4;25(1):452. doi: 10.1186/s13063-024-08294-4. PMID 38965542
- See also: Initial trial registration published under embargo — http://osf.io/46twc